CLINICAL TRIAL: NCT06509074
Title: Beta-Blockers in Takotsubo Syndrome Study: A Randomized Clinical Trial (β-Tako)
Brief Title: Beta-Blockers in Takotsubo Syndrome Study
Acronym: β-Tako
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Fernando Alfonso, Head Cardiac Department, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Takotsubo Cardiomyopathy; Beta-blockers; Echocardiography; Left Ventricular Function
Keywords: Takotsubo Cardiomyopathy; beta-blockers; echocardiography; left ventricular function; acute myocardial infarction; acute coronary syndrome; coronary angiography; Normal coronary arteries; Heart failure; stress
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Acute Coronary Syndrome; Heart Failure | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: Randomized trial with 2 arms
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors blinded to treatment allocation Blinded independent clinical event committee PROBE initiative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-blockers (Experimental): Beta-blockers with alpha or NO activity will be used. Dosage according to responsible physician and current clinical practice
  Interventions: Drug: Beta blocker
- No beta-blockers (No Intervention): No beta-blockers

INTERVENTIONS:
Drug: Beta blocker — Pragmatic design. Any beta-blocker with alpha or NO activity may be used
  Other Names: Other medications according to local clinical practice protocols and current guidelines
  Arms: Beta-blockers

SUMMARY:
The Beta-blockers in Takotsubo syndrome (TTS) (β-Tako) trial, is an academic, pragmatic, prospective, multicenter randomized clinical trial, aiming to assess the efficacy of beta-blockers (BB) in TTS patients. Two-hundred patients with TTS will be randomized (1:1) to BB (n=100) or no BB (n=100). BB with alpha or nitric oxide release activity will be used in the treatment arm. The primary endpoint will be the comparison of the wall motion score index by echocardiography at 7 days. A composite clinical endpoint (death, stroke, admission for recurrent TTS, ACS, heart failure or atrial fibrillation) at 1 year, will be assessed by an independent clinical events committee. Several sub-studies will be performed. The β-Tako trial will inform treatment decisions in this uniquely challenging clinical entity.

DETAILED DESCRIPTION:
Takotsubo syndrome (TTS) is a cardiac condition mimicking acute coronary syndrome (ACS), characterized by transient left ventricular (LV) dysfunction in the presence of normal coronary arteries. Its etiology remains unknown but reversible microvascular dysfunction secondary to an adrenergic surge appears implicated. Treatment is empiric although in clinical practice most patients receive beta-blockers (BB). The Beta-blockers in TTS (β-Tako) trial, is an academic, pragmatic, prospective, multicenter randomized clinical trial, aiming to assess the efficacy of BB in TTS patients. TTS diagnosis will be confirmed by invasive coronary angiography and serial echocardiographic studies. Two-hundred patients with TTS will be randomized (1:1) to BB (n=100) or no BB (n=100). BB with alpha or nitric oxide release activity will be used in the treatment arm. The primary endpoint will be the comparison of the wall motion score index by echocardiography at 7 days, analyzed in an independent corelab. Changes in LV ejection fraction and global longitudinal strain will be also evaluated. A composite clinical endpoint (death, stroke, admission for recurrent TTS, ACS, heart failure or atrial fibrillation) at 1 year, will be assessed by an independent clinical events committee. Several sub-studies (clinical, imaging, biomarkers, pharmacogenetic, mRNAs, quality of life) will be performed. The β-Tako trial will generate valuable scientific evidence to address unmet clinical needs and inform clinical and treatment decisions in this uniquely challenging clinical entity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Diagnosis of TTS with exclusion of significant coronary artery disease (CAD) by invasive coronary angiography

Exclusion Criteria:

* Patients diagnosed of TTS > 48 hours before.
* Persistent ccardiogenic shock or severe hemodynamic instability
* Persistent severe (>30 mmHg) intraventricular gradient
* Previous diagnosis of severe valvular or ventricular disease or prior myocardial infarction secondary to atherosclerotic CAD
* Patients already receiving treatment with betablockers (*)
* Absolute contraindication/indication for beta-blockers (**)
* Poor echocardiographic window
* Pregnant or breastfeeding women.
* Participation in another clinical trial.

(*) Betablockers at a therapeutic dose at the time of symptom´s onset. (**) Close ECG monitoring required in patients with hypotension, bradycardia or cQT interval prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wall motion score index | 7 days
  Wall motion score index by echocardiography to assess recovery of left ventricular function Wall motion score index (WMSI) ranges from 1 to 4 (1 is normal and 4 worse)

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 7 days
  Left ventricular ejection fraction by echocardiography to assess recovery of left ventricular function
Global longitudinal strain | 7 days
  Global longitudinal strain by echocardiography to assess recovery of left ventricular function
Delta (Change) in: wall motion score index, left ventricular ejection fraction, global longitudinal strain | 7 days
  Changes in LV function by imaging
Delta (Change) in: wall motion score index, left ventricular ejection fraction, global longitudinal strain | 1 month
  Changes in LV function by imaging
Combined clinical endpoint (death, stroke, recurrent TTS, heart failure, acute coronary syndrome, atrial fibrillation | 1 year
  Combined clinical endpoint
Individual endpoints of the combined clinical endpoint Occurrence of death, stroke, recurrent TT, heart failure, acute coronary syndrome, atrial fibrillation will be analyzed and compared individually | 1 year
  Individual clinical endpoints Occurrence of death, stroke, recurrent TT, heart failure, acute coronary syndrome, atrial fibrillation will be analyzed and compared individually in the 2 groups
Angina and quality of life status during daily life assessed in routine clinical practice | 1 year
  Evaluated in clinical visits

OTHER OUTCOMES:
Cardiac Magnetic Resonance (CMR) | 1 year
  CMR to detect edema, late gadolinium enhancement to correlate with clinical data and prognosis
ECG | 1 year
  Correlation of ECG findings with clinical features and prognosis Different ECG parameters will be correlated with the echocardiographic and clinical outcome measures to detect potential correlations
Pharmacogenetic substudy | 1 year
  To assess pharmacogenetic implications of different beta-blockers used The pharcacogenetics of the 2 different betablockers used in this study will be studied in relation to the main echocardiographic and clinical endpoints
Coronary angiography | 1 year
  To assess correlation with angiographic features and clinical findings and prognosis
Biomarkers, inflammatory data, mRNAs | 1 year
  Association with clinical findings and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Alfonso, MD, Study Chair — Hospital Universitario La Princesa, Madrid. IIS-IP
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be considered to be shared by the PI and steering committee, upon adequate and justified request, within a defined scientific research project, and providing adequate supervision of the analysis and credit to the original inverstigators is prearranged
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after publication of the main combined clinical endpoint
Access Criteria: to be defined

REFERENCES:
- [Derived] Alfonso F, Salamanca J, Nunez-Gil I, Ibanez B, Sanchis J, Sabate M, Velazquez M, Raposeiras-Roubin S, Garcia-Camarero T, Antuna P, Mejia H, Carrillo X, Buera I, Martinez-Selles M, Escudier-Villa JM, Sanchez-Prieto J, Blanco Ponce E, Cabezon G, Fernandez-Golfin C, Pascual-Figal D, Cid B, Marcano A, Gonzalez-Manzanares R, Jimenez-Valero S, Vazquez JM, Sanz-Sanchez J, Cecconi A, Del Val D, Abad-Santos F, Crea F. Rationale and design of the beta-blockers in tako-tsubo syndrome study: a randomized clinical trial (beta-Tako). Rev Esp Cardiol (Engl Ed). 2025 Jul;78(7):592-599. doi: 10.1016/j.rec.2024.12.006. Epub 2024 Dec 30. English, Spanish. PMID 39743172